CLINICAL TRIAL: NCT02240927
Title: Comparison of Different Anticoagulation Regimens in Pregnant Patients With Prosthetic Heart Valves: A Randomized Clinical Trial
Brief Title: Anticoagulation Regimens in Pregnant Patients With Prosthetic Heart Valves
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, MEHMET OZKAN, Principal Investigator, MD., Prof., Head of Cardiology, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOSUYOLU1
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Pregnancy; Heart; Complications, Valve, Prosthesis
Keywords: Anticoagulation; Prosthetic Heart Valves; Pregnancy; Warfarin; Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — Enoxaparin; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Enoxaparine (Active Comparator): During first trimester, warfarin is stopped and enoxaparine is started in 1mg/kg dose twice a day. Dose is adjusted according to Anti Factor Xa levels (between 0.7-1.2). Full dose warfarin is continued after first trimester and dose is regulated according to INR level (between 2.5-4).
  Interventions: Drug: Low Molecular Weight Heparine : Enoxaparine
- Enoxaparine and 2.5 mg warfarin (Active Comparator): If the patient's therapeutic warfarin dose is more than 5 mg before pregnancy, warfarin dose is decreased to 2.5 mg during the first trimester and combined with enoxaparine in 1mg/kg dose twice a day. Enoxaparine dose is adjusted according to anti-factor Xa levels (between 0.5-1.0). Full dose warfarin is continued after first trimester and dose is regulated according to INR (between 2.5-4)
  Interventions: Drug: Enoxaparine and 2.5 mg Warfarin
- Enoxaparine and 4 mg warfarin (Active Comparator): If the patient's warfarin consumption dose is more than 5 mg before pregnancy, warfarin dose is decreased to 4 mg during the first trimester and combined with enoxaparine in 1mg/kg dose twice a day. Enoxaparine dose is adjusted according to anti-factor Xa levels (between 0.5-1). Full dose warfarin is continued after first trimester and dose is regulated according to INR level (between 2.5-4).
  Interventions: Drug: Enoxaparine and 4mg Warfarin
- Warfarin (Active Comparator): If the patient's therapeutic warfarin dose is less than 5 mg before pregnancy, warfarin is continued in the same dose during all the pregnancy and the dose is adjusted according to INR level (between 2.5-4).
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Low Molecular Weight Heparine : Enoxaparine — During first trimester, warfarin is stopped and enoxaparine is started in 1mg/kg dose twice a day. Dose is adjusted according to Anti Factor Xa levels (between 0.7-1.2). Full dose warfarin is continued after first trimester and dose is regulated according to INR level (between 2.5-4).
  Other Names: Clexane
  Arms: Enoxaparine
Drug: Enoxaparine and 2.5 mg Warfarin — If the patient's therapeutic warfarin dose is more than 5 mg before pregnancy, warfarin dose is decreased to 2.5 mg during the first trimester and combined with enoxaparine in 1mg/kg dose twice a day. Enoxaparine dose is adjusted according to anti-factor Xa levels (between 0.5-1). Full dose warfarin is continued after first trimester and dose is regulated according to INR level (between 2.5-4)
  Other Names: Clexane and 2.5 mg Warfarin
  Arms: Enoxaparine and 2.5 mg warfarin
Drug: Enoxaparine and 4mg Warfarin — If the patient's warfarin consumption dose is more than 5 mg before pregnancy, warfarin dose is decreased to 4 mg during the first trimester and combined with enoxaparine in 1mg/kg dose twice a day. Enoxaparine dose is adjusted according to anti-factor Xa levels (between 0.5-1). Full dose warfarin is continued after first trimester and dose is regulated according to INR level (between 2.5-4).
  Other Names: Clexane and 4 mg Warfarin
  Arms: Enoxaparine and 4 mg warfarin
Drug: Warfarin — If the patient's therapeutic warfarin dose is less than 5 mg before pregnancy, warfarin is continued in the same dose during all the pregnancy and the dose is adjusted according to INR level (between 2.5-4).
  Arms: Warfarin

SUMMARY:
Pregnancy is associated with increased risk of thrombosis among women with mechanical prosthetic heart valves.However, the best anticoagulant treatment strategies for pregnant patients with prosthetic heart valves have been controversial. In this study the investigators wanted to identify the most effective and safe regimen among different anticoagulant regimens.

DETAILED DESCRIPTION:
Four different anticoagulant treatment regimens for pregnant patients with prosthetic heart valves have been described. In the first arm warfarin is stopped and enoxaparine is started in 1mg/kg dose twice a day which is monitored by weekly anti-Xa levels (between 0.7-1.2) during the first trimester and followed by only warfarin after first trimester. In the second arm, if the patient's warfarin consumption is more than 5 mg before pregnancy, warfarin dose is decreased to 2.5 mg during the first trimester combined with enoxaparine in 1mg/kg dose twice a day; adjusted by measurements of anti-Xa levels (between 0.5-1) weekly until the end of 12th week of pregnancy . In the third arm warfarin dose is decreased to 4 mg during the first trimester combined with enoxaparine given in a similar manner. If the patient's therapeutic warfarin dose is less than 5 mg before pregnancy, warfarin is continued in the same dose during all the pregnancy in the 4th arm. All patients are followed by serial transesophageal echocardiography performed at 0,3,6 and 9. months of pregnancy. Informed consent is taken from all patients. After delivery the babies are examined by a experinced pediatrician and pediatric cardiologist for any congenital anomalies.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients with prosthetic heart valves

Exclusion Criteria:

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Successful pregnancy | 12 month
  In the absence of fetal and maternal fatal or nonfatal major complications successful pregnancy
Maternal Complications | Participants will be followed during pregnancy and postpartum period, an expected average of 12 months
  * Nonfatal major complication: Ischemic stroke, intracranial hemorrhage, embolism (coronary or peripheral), bleeding requiring transfusion, abortus, placental hemorrhage, Assessment of an increase in thrombus burden more than 50% and/or progression of PVT obstruction by transesophageal echocardiography.
  * Nonfatal minor complication: Bleeding without need for transfusion, TIA.
Fetal Complications | 12 months
  Any congenital anomalia which may be attributed to warfarin or enoxaparine usage during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Ozkan, Prof, Principal Investigator — Kosuyolu Kartal Heart Training and Research Hospital
Locations (1):
- Kosuyolu Kartal Heart Training and Research Hospital, Istanbul, Turkey (Türkiye)